CLINICAL TRIAL: NCT00930449
Title: Effects Of A Computerized Working Memory Training Program On Attention, Working Memory, And Academics, In Adolescents With Severe ADHD/LD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Children's Hospital of Eastern Ontario (Other)
Responsible Party: Principal Investigator, Rosemary Tannock, Senior Scientist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1000013779
Record Dates: First submitted 2009-06-29; First posted 2009-06-30 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Attention Deficit Disorder With Hyperactivity; Learning Disorders
Keywords: Pediatrics; Attention-Deficit Hyperactivity Disorder; Learning Disorder; Computerized Working Memory Training Program
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Learning Disabilities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cogmed Working Memory Training Program (Experimental)
  Interventions: Other: Cogmed Working Memory Training Program.
- Academy of Math® program (Active Comparator)
  Interventions: Other: Academy of Math
- Special Education/Individualized Tutoring (Active Comparator)
  Interventions: Other: Special Education/Individualized Tutoring

INTERVENTIONS:
Other: Cogmed Working Memory Training Program. — This program includes a set of visual-spatial and auditory-verbal WM tasks presented via the computer (see Appendix 1 for a description of these tasks). All tasks involve: a) maintenance of simultaneous mental representations of multiple stimuli; b) unique sequencing of stimulus order in each trial; and c) progressive adaptation of difficulty level as a function of individual performance.
  Training will require about 30 minutes per day, 5 days per week, for 5-6 weeks: participants are required to complete 90 WM trials on each training day. Training plans are individualized and are modified according to performance, but the typical plan includes 13 tasks, with 15 trials of 8 tasks each day.
  Arms: Cogmed Working Memory Training Program
Other: Academy of Math — This is an established evidence-based program designed to help at-risk learners (Grades K-12) develop mathematical proficiency by incorporating a mastery-learning approach to foster conceptual understanding, computational fluency, and strategic competency across 10 mathematical subject areas.
  Training is will require about 30 minutes, 5 days per week, for the same duration as the WM program (5-6 weeks), with a counselor or teacher acting as the training aide.
  Arms: Academy of Math® program
Other: Special Education/Individualized Tutoring — Students in this group will receive an additional 30 minutes daily of individualized supplemental instruction in their area of greatest academic need.
  Arms: Special Education/Individualized Tutoring

SUMMARY:
Our primary aim is to determine whether a computerized working memory (WM) training program will help students with severe learning and attention problems, in terms of improving their WM. Additional aims are to determine whether the WM training will also result in improvements in the students' concentration and school work, and how long any beneficial effects will last (i.e., whether the students will continue to show improvements once the training program has stopped).

DETAILED DESCRIPTION:
We have established a collaborative partnership between OISE, HSC, OPDS, and JVS to evaluate the effectiveness of a WM training program when conducted in a school setting. To determine whether the WM training program does improve WM, attention, behaviour, and/or academic achievement, we will compare its effects to those expected to result from two other intervention programs that focus on academic skills only: 1) a computerized software program known to improve math skills (Academy of Math®); and 2) extra, individualized tutoring in an area of academic weakness supervised by a trained and experienced staff person. We will assess WM, related cognitive abilities, ADHD symptoms, academic achievement, before and after intervention, and also at 3- and 6-month follow-up to determine whether any improvements are sustained and increased after the training has finished.

ELIGIBILITY:
Inclusion Criteria:

* fulltime enrollment at one of the three English-language speaking OPDS schools
* confirmed diagnosis of a specific LD with or without comorbid ADHD
* IQ > 80 (based on WISC-IV)
* English as the primary spoken language

Exclusion Criteria:

* uncorrected sensory impairments (vision, hearing)
* severe comorbid mental health disorders requiring medications other than those used for ADHD or intensive treatment
* severe impairments in oral communication, impeding intelligibility of spoken responses

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2008-11; Primary Completion 2011-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
CANTAB Spatial Working Memory | 15-20 min
Automated Working Memory Assessment Listening Recall | 15-20 min

SECONDARY OUTCOMES:
Teacher - Strengths and Weakness of ADHD-symptoms and Normal-behavior scale (SWAN) | 5 min/student
Teacher - Children's Organizational Skills Scale | 5 min/student
Wide Range Achievement Test 4 Progress Monitoring Version: word reading, spelling, sentence comprehension, math computation | 10-15 min

CONTACTS AND LOCATIONS:
Overall Officials: Rosemary Tannock, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (2):
- Canada (2):
  - Ontario Provincial and Demonstration Schools, Milton, Ontario
  - The Hospital for Sick Children, Toronto, Ontario